CLINICAL TRIAL: NCT01778127
Title: A Randomized Web-Based Physical Activity Intervention in Adolescent Survivors of Childhood Cancer
Brief Title: A Web-Based Physical Activity Intervention in Adolescent Survivors of Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ZAMZEE; NCI-2013-00384 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: Cancer Survivor; Physical Activity; Health Outcomes; Rewards-Based Intervention; Cardiovascular Health; Musculoskeletal Health; Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A: Minimal Rewards (Experimental): Participants use an activity monitor and the interactive website. They will receive minimal rewards based on their physical activity levels.
  Interventions: Behavioral: Activity Monitor; Behavioral: Interactive Website; Behavioral: Educational Materials
- Group B: Immediate Incentives (Experimental): Participants use an activity monitor and the interactive website.
  In addition to minimal rewards, participants will receive immediate incentives as they move from one level to the other on the website.
  Interventions: Behavioral: Activity Monitor; Behavioral: Interactive Website; Behavioral: Educational Materials
- Group C: Control (Experimental): Participants in the control group will receive an activity monitor and educational materials, but will not have access to the interactive website. No rewards will be offered for their participation.
  Interventions: Behavioral: Activity Monitor; Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Activity Monitor — Measurement of physical activity.
  Other Names: Tri-Axial Accelerometer; Zamzee
Behavioral: Interactive Website — Zamzee is a meter that measures activity and a website that makes moving fun. Parents of participants can set activity goals. Activity is uploaded to the website where participants track progress and earn rewards by increasing their level of activity. Participants can view leaderboards and check how other participants are doing.
  Other Names: Zamzee Website
  Arms: Group A: Minimal Rewards; Group B: Immediate Incentives
Behavioral: Educational Materials — All participants will receive educational handouts about physical activity. Participants will receive the educational handouts again via mail three and five months into the study to reinforce the importance of physical activity and maintain compliance.
  Other Names: Educational Brochure

SUMMARY:
Five year survival following a diagnosis of childhood cancer has reached 83%, making long term health outcomes among survivors an important concern. The growing population of survivors is at an increased risk of physical inactivity and associated adverse health outcomes. Regular physical activity is associated with better cardiovascular and musculoskeletal health. Despite the known benefits of physical activity, nearly half of all childhood cancer survivors do not meet recommended guidelines for physical activity.

Researchers at St. Jude Children's Research Hospital (SJCRH) want to determine if a rewards-based physical activity intervention delivered via an interactive website among young adolescent childhood cancer survivors, aged 11 through 14 years, will increase physical activity levels and improve cardiovascular and musculoskeletal health. The investigators also want to learn if this rewards-based intervention is effective. To achieve this goal the investigators have designed a three-arm prospective, randomized study with two reward-based intervention groups and a control group.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* To compare changes in levels of moderate and vigorous physical activity over 24 weeks.

SECONDARY OBJECTIVE:

* To compare changes in cardiorespiratory fitness, muscular strength and flexibility over 24 weeks.

Participants will be randomized to one of three groups. Participants in the control group will receive an activity monitor and educational materials, but will not have access to the interactive website. Participants randomized to the two intervention groups will be given access to a rewards program delivered via an interactive website, an activity monitor, and educational materials. Individual physical activity data can be viewed by study participants after uploading information from their monitors to the interactive website. One intervention group will receive minimal rewards, while the other group will receive immediate incentives as well as the minimal rewards as they move from one level to the other on the website.

After 24 weeks, changes in cardiorespiratory fitness, muscular strength, flexibility, and physical function will be compared between the two intervention groups and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated for childhood cancer at St. Jude Children's Research Hospital (SJCRH)
* 11 through 14 years of age
* Not undergoing active treatment for cancer
* Medical clearance from participant's attending physician via email
* Does not meet the Centers for Disease Control (CDC) physical activity guidelines. CDC guidelines for children age 11 to 14 are defined as 60 minutes or more per day of physical activity, seven days a week
* Internet access and a computer that has software that is compatible with the study device (Windows XP, Windows Vista, Windows 7, Mac OSX 10.5 and Mac OSX 10.6)

Exclusion Criteria:

* Global cognitive impairment (Full Scale Intelligence Quotient < 70) that prevents use of the interactive website
* Pregnant female
* Inability to read and write English

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K. Ness, PT, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol enrolled 105 participants at St. Jude Children's Research Hospital from 9/2013 through 4/2014. Of the 105, 5 were determined to be ineligible after baseline screening (4 too active; 1 did not meet IQ criteria), and 2 withdrew prior to randomization but after baseline testing. The remaining 98 were randomized.
Pre-assignment Details: 98 participants were randomized 1:1:1 stratified by gender into 3 groups. Randomization was implemented using software based on Zelen's methodology. The principal investigator and study staff were blind to group assignment.
Groups:
- Group B: Immediate Incentives: Participants use an activity monitor and the interactive website.
  In addition to minimal rewards, participants will receive immediate incentives as they move from one level to the other on the website.
  Activity Monitor: Measurement of physical activity.
  Interactive Website: Zamzee is a meter that measures activity and a website that makes moving fun. Parents of participants can set activity goals. Activity is uploaded to the website where participants track progress and earn rewards by increasing their level of activity. Participants can view leaderboards and check how other participants are doing.
  Educational Materials: All participants will receive educational handouts about physical activity. Participants will receive the educational handouts again via mail three and five months into the study to reinforce the importance of physical activity and maintain compliance.
Period: Overall Study
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Started | 33 | 33 | 32
Completed | 25 | 31 | 26
Not Completed | 8 | 2 | 6
Not completed — Lost to Follow-up | 5 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control | Total
Number analyzed (Participants) | 25 | 31 | 26 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (1.2) | 12.8 (0.9) | 12.6 (1.2) | 12.8 (1.1)
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at diagnosis | 3.0 (3.1) | 4.2 (3.0) | 3.6 (2.5) | 3.6 (2.9)
  Time since diagnosis | 10.0 (3.0) | 8.6 (3.1) | 9.0 (2.7) | 9.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 14 | 44
  Male | 11 | 15 | 12 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Non-White | 3 | 6 | 8 | 17
  White | 22 | 25 | 18 | 65
Diagnosis [Number; unit: participants]
  Leukemia | 5 | 7 | 7 | 19
  Central Nervous System Tumor | 7 | 7 | 4 | 18
  Lymphoma | 2 | 2 | 4 | 8
  Retinoblastoma | 6 | 5 | 2 | 13
  Other Solid Tumor | 5 | 10 | 9 | 24
Daily Moderate to Vigorous Physical Activity (MVPA) [Mean (Standard Deviation); unit: minutes] | 26.8 (15.7) | 28.0 (16.6) | 32.3 (22.6) | 29.0 (18.2)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (6.6) | 22.6 (6.3) | 22.8 (5.5) | 23.4 (6.1)
Resting heart rate (HR) [Mean (Standard Deviation); unit: beats/minute] | 82.8 (11.2) | 80.4 (14.5) | 81.5 (14.9) | 81.5 (13.6)
Resting respiratory rate (RR) [Mean (Standard Deviation); unit: breaths/minute] | 19.2 (1.1) | 19.0 (1.3) | 18.4 (1.7) | 18.9 (1.4)
Blood pressure (BP) [Mean (Standard Deviation); unit: mmHG]
  Systolic | 115.6 (9.8) | 113.5 (9.9) | 117.6 (11.2) | 115.4 (10.3)
  Diastolic | 68.2 (7.3) | 66.2 (7.2) | 68.5 (9.3) | 67.5 (7.9)
Peak VO2 [Mean (Standard Deviation); unit: ml/kg/min] — Peak VO2 is a measure of exercise capacity: volume of oxygen uptake per minute adjusted for weight.
  ml/kg/min | 30.0 (7.9) | 30.0 (7.8) | 31.2 (6.6) | 30.4 (7.5)
Sit and reach [Mean (Standard Deviation); unit: cm] — Sit and reach is a measure of low back and hamstring flexibility.
  cm | 21.7 (8.9) | 19.6 (9.8) | 22.2 (10.4) | 21.1 (9.7)
Active dorsiflexion [Mean (Standard Deviation); unit: degrees] — Active dorsiflexion is a measure of ankle flexibility.
  degrees | 13.1 (7.6) | 13.6 (8.1) | 14.3 (8.6) | 13.7 (8.1)
Hand grip [Mean (Standard Deviation); unit: kg] — Hand grip is a measure of how much muscle power a person can generate gripping an object.
  kg | 20.9 (6.3) | 19.0 (5.6) | 22.5 (7.1) | 20.7 (6.3)
Sit-up [Mean (Standard Deviation); unit: sit-ups] — This measure assessed the number of sit-ups done in 30 seconds.
  sit-ups | 14.3 (5.1) | 15.2 (6.1) | 16.2 (6.2) | 15.2 (5.8)
Pushup [Mean (Standard Deviation); unit: push-ups] — This measure assessed the number of push-ups done in 30 seconds.
  push-ups | 9.6 (6.6) | 13.3 (5.9) | 12.4 (7.5) | 11.9 (6.6)
Quadriceps [Mean (Standard Deviation); unit: Newton meters (Nm)/kg]
  at 60 degrees/second | 156.3 (46.0) | 164.2 (46.3) | 159.9 (41.0) | 160.4 (44.5)
  at 120 degrees/second | 136.5 (36.2) | 142.0 (41.7) | 137.8 (36.5) | 139.0 (38.4)
  at 180 degrees/second | 117.6 (32.9) | 121.7 (36.7) | 118.6 (29.5) | 119.4 (33.3)
Dorsiflexion [Mean (Standard Deviation); unit: Nm/kg]
  at 30 degrees/second | 21.7 (8.7) | 26.5 (14.9) | 27.9 (15.0) | 25.5 (13.0)
  at 60 degrees/second | 19.9 (7.4) | 24.7 (12.0) | 25.5 (11.1) | 23.5 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Differences in Change in Daily Average of Moderate and Vigorous Physical Activity (MVPA) Levels Between Groups
Description: The impact of the intervention was assessed at the end of 24 weeks by comparing the mean difference in physical activity levels from baseline to 24-weeks between groups.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
minutes | -2.58 (13.70) | -2.12 (12.95) | -7.78 (13.70)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.90, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.18, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.14, t-test, 2 sided

2. Secondary Outcome: Differences in Change in Cardiovascular Function Between Groups Over 24 Weeks
Description: The difference in mean change in peak oxygen uptake from baseline to 24-weeks was compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
ml/kg/min | -0.21 (5.15) | -1.19 (4.70) | 0.09 (5.25)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.49, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.84, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.37, t-test, 2 sided

3. Secondary Outcome: Differences in Change in Flexibility Between Groups Over 24 Weeks: Sit and Reach
Description: The difference in mean changes of sit and reach from baseline to 24-weeks was compared between groups
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
cm | -0.71 (4.85) | 2.25 (4.50) | -0.02 (4.85)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.63, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.09, t-test, 2 sided

4. Secondary Outcome: Differences in Change in Flexibility Between Groups Over 24 Weeks: Active Dorsiflexion
Description: The difference between mean changes from baseline to 24-weeks in active dorsiflexion was compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
degrees | -1.72 (6.40) | -0.55 (5.70) | -0.32 (6.25)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.49, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.43, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.89, t-test, 2 sided

5. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Hand Grip
Description: The difference from baseline to 24-weeks in mean changes in grip strength (kilograms) was compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
kg | 1.47 (3.50) | 0.98 (3.20) | 1.00 (3.45)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.61, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.64, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.99, t-test, 2 sided

6. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Sit-up
Description: The number of sit-ups completed in 30 seconds was assessed, and the differences from baseline to 24-weeks in mean changes on the strength subtests of the Bruininks-Oseretsky Test of Motor Proficiency were compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Sit-ups
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
Sit-ups | 2.67 (5.65) | 3.29 (5.25) | 2.43 (5.80)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.69, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.89, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.59, t-test, 2 sided

7. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Pushup
Description: The number of push-ups completed in 30 seconds was assessed, and the differences from baseline to 24-weeks in mean changes on the strength subtests of the Bruininks-Oseretsky Test of Motor Proficiency were compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Pushups
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
Pushups | 2.37 (5.70) | 1.93 (5.40) | 2.27 (5.95)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.78, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.95, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.83, t-test, 2 sided

8. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Quadriceps at 60 Degrees/Second
Description: The difference from baseline to 24-weeks in mean changes in knee extension strength 60 degrees per second (Newton meters) was compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Newton meters (Nm)/kg
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
Newton meters (Nm)/kg | -4.10 (34.80) | -2.05 (31.55) | -1.91 (34.80)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.83, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.83, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.99, t-test, 2 sided

9. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Quadriceps at 120 Degrees/Second
Description: The difference from baseline to 24-weeks in mean changes in knee extension strength 120 degrees per second (Newton meters) was compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
Nm/kg | -6.62 (28.95) | -0.59 (25.70) | 4.16 (28.35)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.44, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.19, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.54, t-test, 2 sided

10. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Quadriceps at 180 Degrees/Second
Description: The difference from baseline to 24-weeks in mean changes in knee extension strength at 180 degrees per second (Newton meters) was compared between groups
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
Nm/kg | -0.64 (28.10) | 0.78 (25.50) | 2.55 (28.10)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.17, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.13, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.81, t-test, 2 sided

11. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Dorsiflexion at 30 Degrees/Second
Description: The differences from baseline to 24-weeks in mean changes in ankle dorsiflexion strength 30 degrees per second (Newton meters) was compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
Nm/kg | 3.94 (16.25) | -3.74 (14.75) | -2.81 (16.65)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.08, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.15, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.83, t-test, 2 sided

12. Secondary Outcome: Differences in Change in Muscular Strength Between Groups Over 24 Weeks: Dorsiflexion at 60 Degrees/Second
Description: The differences from baseline to 24-weeks in mean changes in ankle dorsiflexion strength at 60 degrees per second (Newton meters) was compared between groups.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Number analyzed (Participants) | 25 | 31 | 26
Nm/kg | 3.82 (12.85) | -3.00 (11.65) | -2.14 (13.15)
Statistical Analysis 1: Comparison: Group A: Minimal Rewards vs Group B: Immediate Incentives; Test type: Superiority or Other; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: Minimal Rewards vs Group C: Control; Test type: Superiority or Other; p = 0.11, t-test, 2 sided
Statistical Analysis 3: Comparison: Group B: Immediate Incentives vs Group C: Control; Test type: Superiority or Other; p = 0.81, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the on-study date until the completion of the intervention up to 24 weeks later.
Arm/Group | Group A: Minimal Rewards | Group B: Immediate Incentives | Group C: Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/31 | 0/26
Other Adverse Events (participants affected / at risk) | 2/25 | 0/31 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Minimal Rewards (N=25) | Group B: Immediate Incentives (N=31) | Group C: Control (N=26)
Abnormal ECG (Cardiac disorders) | 2 (25) | 0 (0) | 0 (0) — Two children had abnormal ECG findings on their baseline cardiopulmonary fitness tests and were referred to their primary care physician. Neither was related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes